CLINICAL TRIAL: NCT05507619
Title: Heat and Acupuncture Randomised Controlled Trial to Manage Osteoarthritis of the Knee (HARMOKnee)
Brief Title: Heat and Acupuncture Randomised Controlled Trial to Manage Osteoarthritis of the Knee
Acronym: HARMOKnee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: National Healthcare Group, Singapore (Other Government); Singapore Chung Hwa Medical Institution (Other)
Responsible Party: Principal Investigator, Bryan Tan, Consultant, National Healthcare Group, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/01106
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy; Diathermy; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Other: Standard Care
- Intervention (Experimental)
  Interventions: Other: Acupuncture with Heat Therapy + Standard Care

INTERVENTIONS:
Other: Acupuncture with Heat Therapy + Standard Care — Biweekly sessions of acupuncture with heat therapy over 6 weeks (total 12 sessions), in addition to standard care (e.g. physiotherapy, dietetics, pain management).
  Arms: Intervention
Other: Standard Care — Treatment as prescribed by orthopaedic surgeon routinely (e.g. physiotherapy, dietetics, pain management)
  Arms: Control

SUMMARY:
Knee osteoarthritis (KOA) is one of the largest and fast-growing causes of pain, impaired mobility, and poor quality of life in the elderly worldwide. Despite a significant increase in Traditional Chinese Medicine (TCM) utilisation, in particular acupuncture, as first or second-line treatment among local KOA patients, there exists a lack of high-quality evidence on its efficacy and local practice guidelines for TCM use in KOA tailored to our specific population demographic.

HarmoKNEE trial aims to address these gaps by evaluating the short and medium-term clinical and cost-effectiveness of TCM acupuncture with far-infrared heat therapy in addition to standard care, compared to standard care alone. Through a robust process and economic evaluation, the investigators aim to inform evidence-based practice for KOA patients in Singapore to facilitate the large-scale implementation of a comprehensive and holistic model of care which harmonises elements from Western medicine and TCM.

The investigators hypothesize that acupuncture with heat therapy as an adjunct to standard care is clinically more effective than standard care alone.

This will be a multi-centre pragmatic, parallel-arm, single-blinded, effectiveness-implementation hybrid randomised control trial. KOA patients will be randomised to either the control arm (standard care only) or intervention arm (biweekly sessions of acupuncture with heat therapy over 6 weeks, in addition to standard care).

A mixed-method approach through an embedded process evaluation will facilitate large scale implementation. An economic evaluation will be performed to evaluate financial sustainability

ELIGIBILITY:
Inclusion Criteria:

1. 45 to 99 years old
2. Independent Community Mobilizers with or without walking aids
3. Conversant in English or Chinese
4. NICE clinical criteria for OA knee

Exclusion Criteria:

1. Alternative diagnosis to KOA e.g., referred pain from the spine or hip
2. Other forms of arthritis eg., inflammatory, post-traumatic
3. Inability to comply with study protocol e.g., cognitive impairment
4. Previous knee arthroplasty
5. Wheelchair-bound patients
6. Medical conditions that will medically interfere with study involvement e.g., decompensated heart failure, stroke, end-stage renal failure
7. Allergies to metal (needles)

Ages: 45 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2022-08-17 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Knee Osteoarthritis Outcome Score (KOOS-12) | Baseline, Change from Baseline to 6 weeks, Change from Baseline to 3 months, Change from Baseline to 6 months
  Derived from the original 42-item Knee injury and Osteoarthritis Outcome Score (KOOS), KOOS-12 reduces respondent burden by 70% from the original KOOS while providing scale scores for knee-specific Pain, Function and QOL, along with a summary measure of overall knee impact. The KOOS sub scales are scored using the method of summated ratings and transformed to range from 0 to 100, with 0 representing extreme knee problems and 100 representing no knee problem. The KOOS-12 Summary knee impact score is calculated as the average of the KOOS-12 Pain, KOOS-12 Function and KOOS-12 QOL scale scores. It also ranges from 0 to 100, where 0 is the worst possible and 100 is the best possible score.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcomes Score (KOOS) subscales - Pain, Function, QoL | Baseline, Change from Baseline to 6 weeks, Change from Baseline to 3 months, Change from Baseline to 6 months
  The three subscales of KOOS-12 are scored separately: KOOS Pain (4 items); KOOS Function (4 items); KOOS QoL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the three scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
EuroQol-5 Dimensions (EQ-5D-5L) | Baseline, Change from Baseline to 6 weeks, Change from Baseline to 3 months, Change from Baseline to 6 months
  EuroQol-5 Dimensions (EQ-5D) consists of 2 dimensions, the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by selecting the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS will be used as a quantitative measure of health outcome.
Patient Health Questionnaire 4 (PHQ-4) | Baseline, Change from Baseline to 6 weeks, Change from Baseline to 3 months, Change from Baseline to 6 months
  Measurement for depression and anxiety rated on a 4 point Likert-type scale. 0 refers to 'Not at all', 3 refers 'Nearly everyday'. Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
  Total score ≥3 for first 2 questions suggest anxiety. Total score ≥3 for last 2 questions suggest depression.
Pain, Enjoyment, General Activity Scale (PEG) | Baseline, Change from Baseline to 6 weeks, Change from Baseline to 3 months, Change from Baseline to 6 months
  Measures the pain intensity and interference level using a three-item scale. Scale of 0 to 10 is used for each item. 0 refers 'no pain', 10 refers 'worse pain'. Add the responses to the three questions, then divide by three to get a mean score (out of 10) on overall impact of points.
Functional Assessment - 30s chair stand test | Baseline, Change from Baseline to 3 months, Change from Baseline to 6 months
  To test leg strength and endurance. Total number of repetitions completed in 30 seconds is recorded.
Functional Assessment - 40m fast-paced walk test | Baseline, Change from Baseline to 3 months, Change from Baseline to 6 months
  Measure of patient's walking speed. Time taken to complete 40 meters walk will be recorded in seconds.
Functional Assessment - 4 stairs climb test | Baseline, Change from Baseline to 3 months, Change from Baseline to 6 months
  To assess the strength, balance and agility through ascending and descending a set number of steps. Time to ascend and descend steps (excluding turning around time) is recorded separately in seconds. Overall time taken (including the turn around time) to ascend and descend stairs is also recorded.
Functional Assessment - Timed up and go test | Baseline, Change from Baseline to 3 months, Change from Baseline to 6 months
  To assess patient's mobility and balance through the patient's ability to rise from a seated position to walk around a cone 3 meters away and return to the seated position. Time taken to perform the test in fast walking pace will be recorded in seconds.
TCM Evaluation Form | Assess at Week 1 (start of treatment, before the 1st acupuncture session), Week 4 (mid-treatment, before the 7th acupuncture session) and Week 6 (end of treatment, after the 12th / last acupuncture session).
  Used on intervention arm only. Form was designed after considering the progression and severity of KOA defined in TCM clinical guidelines published in China. TCM physician assists to administer the TCM-specific questions.
VAS & ROM Evaluation Form | Assess weekly for the first 6 weeks from the start of treatment
  Used on intervention arm only. Form was designed after considering the progression and severity of KOA defined in TCM clinical guidelines published in China. Assess and completed by attending TCM physician.

OTHER OUTCOMES:
University of California, Los Angeles (UCLA) activity score | Baseline, Change from Baseline to 6 weeks, Change from Baseline to 3 months, Change from Baseline to 6 months
  1 question survey to understands patient physical activity level from a scale of 1 (wholly inactive) to 10 (regular participation in impact sports).
Global perceived effect (GPE) | Assess at 3 months, 6 months, 12 months
  Patient will be asked to rate thier overall recovery on a 7-point Likert scale. 1 refers to 'Very much improved'; 7 refers to 'Very much deteriorated'.
Patient Acceptable Symptom State (PASS) | Assess at 3 months, 6 months, 12 months
  A single-question used to assess patient's satisfaction in the treatment. Response will be either yes or no. "When you think of your knee function, will you consider your current condition as satisfying? By knee function, you should take into account your activities of daily living, sport and recreational activities, your pain and other symptoms and your quality of life."
Self-reported treatment failure | Assess at 3 months, 6 months, 12 months
  Patient who answers 'no' to PASS will be asked to determine if they consider the treatment to have failed. Response will be 'yes' or 'no'. "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?"
Cumulative Analgesia Consumption Score (CACS) | Assess at 3 months, 6 months, 12 months
  Objective measurement of patient's analgesics average weekly consumption based on the quantity multiplied by the category of analgesic medication according to the WHO pain relief ladder (1 point - non-opioid, 2 points - mild opioid, 3 points - strong opioid) in order to calculate a total score.
Questionnaire measuring the direct and indirect costs | Assess at 3 months, 6 months, 12 months
  Cost questionnaire
Adverse Events | Assess at 6 weeks, 3 months, 6 months, 12 months
  Adverse events (AE) and serious adverse events (SAE) will be recorded at all follow-ups by asking the participants about potential AEs using open-probe questioning to ensure that all AEs are recorded. AEs will be categorized into index knee or other sites and will be recorded and assessed for severity independent of whether or not there is a causal relationship with study treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Tan, Principal Investigator — Woodlands Health
Locations (2):
- Singapore (2):
  - Singapore Chung Hwa Medical Institution, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan BY, Tan CY, Tan TL, Yang SY, Chew GLS, Tan SI, Chua YC, Yan YW, Soh DBQ, Goh TH, Ng PJ, Ng YT, Kuan SB, Teo BS, Kong KH, Pereira MJ, Ng HP. Heat and Acupuncture to Manage Osteoarthritis of the Knee (HARMOKnee): Protocol for an Effectiveness-Implementation Hybrid Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 3;13:e54352. doi: 10.2196/54352. PMID 38568718